CLINICAL TRIAL: NCT07269522
Title: Functional Outcomes of Arthroscopic Anterior Cruciate Ligament Reconstruction by Hamstring Graft With and Without Platelet-Rich Plasma
Brief Title: Arthroscopic Anterior Cruciate Ligament Reconstruction by Hamstring Graft With and Without Platelet-Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-NAVEED-LGH
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL reconstruction by hamstring graft with PRP group (Experimental): Patients underwent anterior cruciate ligament reconstruction by hamstring graft along with platelet-rich plasma augmentation applying the standard arthroscopic ACL reconstruction technique.
  Interventions: Procedure: ACL reconstruction by hamstring graft with PRP
- ACL reconstruction by hamstring graft group (Experimental): Patients underwent anterior cruciate ligament reconstruction by hamstring graft without platelet-rich plasma augmentation applying the standard arthroscopic ACL reconstruction technique.
  Interventions: Procedure: ACL reconstruction by hamstring graft

INTERVENTIONS:
Procedure: ACL reconstruction by hamstring graft with PRP — Patients underwent anterior cruciate ligament reconstruction by hamstring graft along with platelet-rich plasma augmentation applying the standard arthroscopic ACL reconstruction technique.
  Arms: ACL reconstruction by hamstring graft with PRP group
Procedure: ACL reconstruction by hamstring graft — Patients underwent anterior cruciate ligament reconstruction by hamstring graft without platelet-rich plasma augmentation applying the standard arthroscopic ACL reconstruction technique.
  Arms: ACL reconstruction by hamstring graft group

SUMMARY:
No local data exists regarding the outcomes of anterior cruciate ligament reconstruction by hamstring graft with and without platelet-rich plasma. This study aimed to compare the functional outcomes of arthroscopic anterior cruciate ligament reconstruction by hamstring graft with and without platelet-rich plasma.

DETAILED DESCRIPTION:
In animal studies, platelet-rich plasma has shown excellent results in accelerating the healing of the anterior cruciate ligament, but studies on human have shown varying clinical outcomes when investigating platelet-rich plasma for its effects on anterior cruciate ligament reconstruction. The findings of this study could provide important insights about the possible role of platelet-rich plasma in arthroscopic anterior cruciate ligament reconstruction by hamstring graft. to enhance early graft healing and reduce early complications, though its long-term effectiveness remains inconsistent. Studies suggest PRP may improve short-to-medium term outcomes like reduced pain and enhanced knee function,

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 18-40 years
* With clinically and radiologically confirmed arthroscopic evidence of ACL injury

Exclusion Criteria:

* With comprised bilateral ACL tears
* Lack of fitness due to associated comorbidity
* Fractures of lower limb bones and/or spine/neurovascular injuries
* Injuries to other knee ligaments
* Significant knee joint arthritis
* Local skin infections

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Anterior Drawer's test | 12 weeks
  Number of patients having grade-1 on the Anterior Drawer's test
Lachman's test | 12 weeks
  Number of patients having grade-1 on the Lysholm knee score
Lysholm knee score | 12 weeks
  A higher Lysholm knee score was labeled as effectiveness of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Ali, FCPS, Principal Investigator — Lahore General Hospital, Lahore, Pakistan; Muhammad Hanif, FCPS, Study Director — Lahore General Hospital, Lahore, Pakistan
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.